CLINICAL TRIAL: NCT05207280
Title: Randomized Clinical Trial Comparing Noradrenaline Plus Placebo Versus Terlipressin Plus Noradrenaline for the Treatment of Septic Shock
Brief Title: Clinical Trial Comparing Noradrenaline (NA) Plus Placebo Versus Noradrenaline Plus Terlipressin (TP) in Septic Shock
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CONTENTSS
Record Dates: First submitted 2021-11-18; First posted 2022-01-26 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Septic Shock
Keywords: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Norepinephrine; Terlipressin

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, multicenter, double-blind clinical trial with two treatment arms
Who Masked: Participant, Investigator
Masking Description: double-blind clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Noradrenaline plus Terlipressin (Experimental): Patients enrolled in this arm, will receive noradrenaline with dose equal to or greater than 0.2 μg / Kg / min for at least 3 hours. Solution for infusion (Intravenous). And: Terlipressin with dose 1 mg every 6 hours diluted in a 50 mL serum to pass in 15-30 minutesin injectable solution. Intravenous (diluted in a 50 mL serum to pass in 15-30 minutes)
  Interventions: Combination Product: Noradrenaline plus Terlipressin
- Noradrenaline plus placebo (Placebo Comparator): Patients enrolled in this arm, will receive noradrenaline with dose equal to or greater than 0.2 μg / Kg / min for at least 3 hours in solution for infusion (Intravenous), and placebo with solution in vial with the same external appearance as terlipressin. 1 mg every 6 hours, diluted in a 50 mL serum to pass in 15-30 minutes in injectable solution Route of administration: Intravenous, diluted in a 50 mL serum to pass in 15-30 minutes
  Interventions: Combination Product: Noradrenaline plus Terlipressin

INTERVENTIONS:
Combination Product: Noradrenaline plus Terlipressin — Comparison Norepinephrine plus placebo versus Terlipressin plus Norepinephrine for the Treatment of Septic Shock
  Other Names: Noradrenaline plus placebo

SUMMARY:
Septic shock is a major health problem. In the clinical practice guidelines of the Surviving Sepsis Campaign is recommended to add vasopressin (VP) or epinephrine in case of not reaching the goal of mean arterial pressure (MAP) although with a low level of evidence.

This is a clinical trial with the purpose of comparing the efficacy and safety of norepinephrine (NE) plus placebo versus NE plus terlipressin (TP) in adult patients with septic shock and with a Sepsis related Organ Failure Assessment score (SOFA)> 4 points. The primary objective will be a combined end-point: reduction of organic dysfunction measured at 72 h by SOFA score and by the increase in ICU (Intensive care unit) -free days measured at 28 days.

DETAILED DESCRIPTION:
Introduction: Septic shock is a major health problem. The clinical practice guidelines of the Surviving Sepsis Campaign establish the use of NE if after resuscitation with fluids a MAP> 65 mm Hg is not achieved. In these guidelines, it is recommended to add VP or epinephrine in case of not reaching the goal of MAP although with a low level of evidence.

TP is a synthetic analogue of VP with a long half-life. Preliminary studies on the use of TP associated with NE have not shown a decrease in mortality, although a reduction in organic dysfunction at 72 h, with discordant data regarding the rate of adverse events.

Material and Methods: Randomized, parallel, double-blind and multicenter clinical trial with the purpose of comparing the efficacy and safety of NE plus placebo versus NE plus TP in adult patients with septic shock and with a SOFA score> 4 points. The threshold dose of NE> 0.2 µg / kg / min is chosen to associate the second vasopressor (TP or placebo). The primary objective will be a combined end-point: reduction of organic dysfunction measured at 72 h by SOFA score and by the increase in ICU -free days measured at 28 days. The secondary objectives will be: mortality at 28 and 90 days, the need of renal replacement therapies, mechanical ventilation-free days, vasopressor-free days, and adverse reactions. Sample size of 152 patients (76 per arm), stratified by center and severity of illness. In addition, 6 single nucleotide polymorphisms of the vasopressin V1a receptor and a polymorphism of leucyl / cystinyl aminopeptidase or vasopressinase will be determined to establish its association with mortality in septic shock and with the efficacy and the occurrence of adverse effects due to the use of TP.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years or older).
2. Patients with septic shock
3. Patients with a SOFA > 4 points.

5. Oxygen saturation in the central venous system > 70% 5. Central venous pressure> 8 mmHg. 6. Signature of the informed consent by the patient or her legal representative.

Exclusion Criteria:

1. Pregnant or lactating patients.
2. Pathologies in which terlipressin is clinically indicated: gastrointestinal bleeding due to esophageal-gastric varices, hepatorenal syndrome.
3. Patients diagnosed with unstable acute coronary syndrome.
4. Patients with acute or chronic mesenteric ischemia.
5. Patients with Raynaud's Phenomenon, or vasospastic disease.
6. Patients participating in another intervention clinical trial.
7. Patients with active bleeding.
8. Patients with renal replacement technique at the time of randomization.
9. Patients with some limitation of life support treatment
10. Previous use of terlipressin during your stay in the intensive Care Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Organ failure | 72 hours
  Number of organ failures related sepsis. Assessment Sepsis related Organ Failure Assessmen scale (SOFA scale) after administration of terlipressin / placebo. These scale assesses organ dysfunction. In patients with infection, a SOFA score ≥ 2 points (in patients with chronic organ dysfunction, a 2 point increase from baseline score) is diagnostic of sepsis.
Days of life free of stay in the Intensive Care Unit | 28 days
  Number of the days of life free of stay in the Intensive Care Unit measured after the administration of terlipressin / placebo

SECONDARY OUTCOMES:
Lactate clearance | 6, 12, 24 and 72 hours
  Measure of the difference between lactate in arterial blood measured at the beginning of vasopressor treatment and that measured at 6, 12, 24 and 72 hours.
Vasopressor-free days of life | 28 days
  Measure of vasopressor-free days of life
Need of renal replacement therapies | 28 days
  Assessment of the change in the need of renal replacement therapies
Mechanical ventilation-free days of life | 28 days
  Measure of days free of mechanical ventilation, by means of the difference between 28 and the sum of the days the patient is under invasive mechanical ventilation or has died.
vasopressor index | 28 days
  Calculation of the vasopressor index, defined as dose of dopamine + dose of dobutamine + dose of epinephrine (x100) + dose of phenylephrine (x100) + dose of terlipressin / placebo.
Mortality | 28 days
  Evaluation of the number of patients who die from the signing of the informed consent until day 28
Mortality | 90 days
  Evaluation of the number of patients who die from the signing of the informed consent until day 90
Adverse effects related to the administration of vasopressors | 90 days
  Measure of the adverse effects related to the administration of vasopressors until the end of study
Relation between organ failure and days of life free of stay in the Intensive Care Unit with the genetic variants of the receptor 1a and LNPEP | 90 days
  Measure of the relation between number of organ failures related sepsis and number of the days of life free of stay in the Intensive Care Unit with the genetic variants of the vasopressin receptor 1a and LNPEP
Relation between the appearance of adverse effects and genetic variants of the receptor 1a and LNPEP. | 90 days
  Measure of the relation between adverse effects due to the use of terlipressin and genetic variants of the vasopressin receptor 1a and LNPEP
Relation of the mortality with genetic variants of the receptor 1a and LNPEP. | 90 days
  Measure of the relation between the mortality with genetic variants of the vasopressin receptor 1a and LNPEP

CONTACTS AND LOCATIONS:
Overall Officials: José Garnacho Montero, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (10):
- Spain (10):
  - Hospital Universitario Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital San Juan de Dios del Aljarafe, Bormujos, Sevilla
  - Hospital Puerta del mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Clínico San Cecilio, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No